CLINICAL TRIAL: NCT00055302
Title: An Open-label Study Evaluating the Safety and Efficacy of Anastrozole™ (ARIMIDEX) in the Treatment of Precocious Puberty in Girls With McCune-Albright Syndrome
Brief Title: Arimidex in McCune Albright Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1033IL/0046; D5394C00046
Record Dates: First submitted 2003-02-25; First posted 2003-02-26 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: McCune-Albright Syndrome
Keywords: vaginal bleeding; advanced bone age; fibrous dysplasia; MAS; McCune-Albright Syndrome
MeSH Terms: conditions — Fibrous Dysplasia, Polyostotic; Uterine Hemorrhage; Fibrous Dysplasia of Bone | interventions — Anastrozole

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Arimidex 1 mg

INTERVENTIONS:
Drug: Arimidex 1 mg — Arimidex (anastrozole) 1mg once daily by mouth

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of anastrozole 1 mg given once daily in subjects with McCune-Albright Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* informed written consent of parent/legal guardian and subject assent (as needed by local requirements)
* females less than or equal to 10 years of age
* diagnosed with McCune-Albright Syndrome
* have progressive precocious puberty

Exclusion Criteria: Any one of the following is regarded as a criterion for exclusion from the study:

* any prior treatment of MAS associated with progressive precocious puberty with a third generation aromatase inhibitor (anastrozole, letrozole, exemestane) in which no clinical response was seen
* concomitant treatment of precocious puberty associated with MAS, with the exception of bisphosphonates for polyostotic fibrous dysplasia and LHRH analogues in the case of central precocious puberty
* liver function tests at screening visit (AST, ALT) > or = 3x the upper limit of the reference range for age
* known hypersensitivity to any component of study medication

Max Age: 10 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2002-08; Primary Completion 2006-02 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The efficacy of study treatment will be assessed based on the change from baseline measurements relating to vaginal bleeding, bone age, and growth velocity | 12 months or until the subject demonstrates the lack of efficacy bases upon progression of primary endpoints or experiences serious drug-related toxicity requiring withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Arimidex Medical Science Director, MD, Study Director — AstraZeneca
Locations (7):
- France (2):
  - Research Site, Montpellier
  - Research Site, Paris
- Germany (3):
  - Research Site, Berlin
  - Research Site, Erlangen
  - Research Site, Osnabrück
- Research Site, Torino, Italy
- Research Site, London, United Kingdom

REFERENCES:
- See also: CSR-1033IL-0046.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1503&filename=CSR-1033IL-0046.pdf